CLINICAL TRIAL: NCT02101021
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of Gemcitabine and Nab-paclitaxel Combined With Momelotinib in Subjects With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma Preceded by a Dose-finding, Lead-in Phase
Brief Title: Gemcitabine and Nab-paclitaxel Combined With Momelotinib in Participants With Previously Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-370-1296; 2014-004480-20 (EudraCT Number)
Record Dates: First submitted 2014-03-28; First posted 2014-04-01 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Momelotinib (Experimental): Participants will receive momelotinib plus nab-paclitaxel and gemcitabine.
  Interventions: Drug: Momelotinib; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Placebo (Placebo Comparator): Participants will receive placebo to match momelotinib plus nab-paclitaxel and gemcitabine.
  Interventions: Drug: Placebo to match momelotinib; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Momelotinib — Tablet (s) administered orally once or twice daily
  Other Names: GS-0387; CYT387
  Arms: Momelotinib
Drug: Placebo to match momelotinib — Placebo to match momelotinib tablets administered orally once or twice daily
  Arms: Placebo
Drug: Nab-paclitaxel — Intravenously administered over approximately 30-40 minutes or as per institutional standard of care on Days 1, 8, and 15 of each cycle
Drug: Gemcitabine — Intravenously administered over approximately 30 minutes or as per institutional standard of care on Days 1, 8, and 15 of each cycle

SUMMARY:
There will be two phases to this study. The lead-in phase will evaluate the safety, pharmacokinetics, and define the maximum tolerated dose (MTD) of momelotinib (MMB) combined with nab-paclitaxel and gemcitabine (nab-P + G) in adults with previously untreated metastatic pancreatic ductal adenocarcinoma. The randomized treatment phase will evaluate the efficacy, safety, and tolerability of nab-P + G with either MMB administered at the MTD or placebo in adults with previously untreated metastatic pancreatic ductal adenocarcinoma. Participants will continue study treatment until disease progression, unacceptable toxicity, consent withdrawal, or participant's refusal of treatment. Following treatment, participants will be followed for safety for 30 days and for survival approximately every 3 months for up to 3 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Presence of metastatic pancreatic adenocarcinoma plus 1 of the following:

  * Histological diagnosis of pancreatic adenocarcinoma confirmed pathologically, OR
  * Pathologist confirmed histological/cytological diagnosis of adenocarcinoma consistent with pancreas origin in conjunction with either:

    * The presence of a mass in the pancreas, OR
    * A history of resected pancreatic adenocarcinoma
* Measurable disease per RECIST v1.1
* Adequate organ function defined as follows:

  * Total bilirubin ≤ 1.25 x upper limit of the normal range (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN
  * Absolute neutrophil count (ANC) > 1500 cells/mm^3, platelet > 100,000 cells/mm^3, hemoglobin > 9 g/dL
  * Serum creatinine < ULN OR calculated creatinine clearance (CrCl) of ≥ 60 ml/min
* Eastern Cooperative Oncology Group (ECOG ) 0 or 1
* Modified Glasgow prognostic score (mGPS) of 1 or 2 at Screening (randomized phase only)

Key Exclusion Criteria:

* Neoadjuvant or adjuvant chemotherapy or chemoradiotherapy for pancreatic adenocarcinoma
* Currently or previously treated with biologic, small molecule, immunotherapy, chemotherapy, or other agents for metastatic pancreatic carcinoma
* Major surgery within 28 days of first dose of study drug
* Minor surgical procedure(s) within 7 days of enrollment or not yet recovered from prior minor surgery (placement of central venous access device, fine needle aspiration, or endoscopic biliary stent ≥ 1 day before enrollment is acceptable)
* Known positive status for HIV
* Chronic active or acute viral hepatitis A, B, or C infection (testing required for hepatitis B and C), or hepatitis B or C carrier
* Peripheral neuropathy ≥ Grade 2
* Known or suspected brain or central nervous system metastases
* Diagnosis of pancreatic islet neoplasm, acinar cell carcinoma, non-adenocarcinoma, adenocarcinoma originating from the biliary tree or cystadenocarcinoma
* History of interstitial pneumonitis and/or require supplemental oxygen therapy
* External biliary drain
* Documented myocardial infarction or unstable/uncontrolled cardiac disease within 6 months of enrollment

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Northwest Medical Specialties, PLLC, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States (US). The first participant was screened on 02 June 2014. The last study visit occurred on 10 April 2017.
Pre-assignment Details: 38 participants were screened.
  Data submitted represent analysis performed on data collected in the lead-in phase by the Study Termination Date, 10 April 2017. The study was discontinued before initiation of the randomized treatment phase, therefore no data were collected for the randomized treatment phase.
Groups:
- MMB Dose Level 1: Momelotinib (MMB) 100 mg tablet once daily + albumin-bound (nab)-paclitaxel plus gemcitabine (nab-P+G) (1000+1000 mg/m^2) intravenous (IV) infusion on Days 1, 8, and 15 of each 28-day cycle
- MMB Dose Level 2: MMB 150 mg tablet once daily + nab-P+G (1000+1000 mg/m^2) IV infusion on Days 1, 8, and 15 of each 28-day cycle
- MMB Dose Level 3: MMB 200 mg tablet once daily + nab-P+G (1000+1000 mg/m^2) IV infusion on Days 1, 8, and 15 of each 28-day cycle
- MMB Dose Level 4: MMB 150 mg tablet twice daily + nab-P+G (1000+1000 mg/m^2) IV infusion on Days 1, 8, and 15 of each 28-day cycle
- MMB Dose Level 5: MMB 200 mg tablet twice daily + nab-P+G (1000+1000 mg/m^2) IV infusion on Days 1, 8, and 15 of each 28-day cycle
Period: Overall Study
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5
Started | 7 | 4 | 7 | 3 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 4 | 7 | 3 | 4
Not completed — Death | 4 | 3 | 6 | 0 | 3
Not completed — Withdrew Consent from study | 1 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All Enrolled Analysis Set: all participants who received a study participant identification number in the study after screening.
Groups:
- MMB Dose Level 1: MMB 100 mg tablet once daily + nab-P+G (1000+1000 mg/m^2) IV infusion on Days 1, 8, and 15 of each 28-day cycle
- Total: Total of all reporting groups
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5 | Total
Number analyzed (Participants) | 7 | 4 | 7 | 3 | 4 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.32) | 63.5 (12.12) | 64.7 (8.79) | 52.0 (5.00) | 59.0 (9.13) | 60.7 (10.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 0 | 1 | 8
  Male | 5 | 1 | 5 | 3 | 3 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  White | 6 | 3 | 6 | 3 | 4 | 22
  Other | 1 | 1 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 4 | 7 | 3 | 4 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 4 | 7 | 3 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Lead-In Phase: Percentage of Participants Experiencing Treatment-Emergent Dose Limiting Toxicity (DLT) Adverse Events
Description: Dose limiting toxicities were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Dose limiting toxicities referred to toxicities experienced during the first 28 days (Cycle 1) of treatment that were judged to be clinically significant and related to study treatment.
  No statistical analysis was planned or performed for this endpoint.
Time Frame: Up to 28 Days
Population: DLT-Evaluable Analysis Set: participants in the Safety Analysis Set who completed all treatment and safety procedures through Day 28, inclusive, or experienced a DLT prior to Day 29. Participants in the DLT-Evaluable Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 3
percentage of participants | 16.7 | 0 | 16.7 | 0 | 0

2. Primary Outcome: Randomized Treatment Phase: Overall Survival (OS)
Description: Overall survival was defined as the time interval from first dose date of MMB to death from any cause
Time Frame: Baseline up to the Date of Death or Censoring, up to 3 years
Population: The study was discontinued before initiation of the randomized treatment phase.
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Lead-In Phase: Overall Survival (OS)
Description: Overall survival was defined as the time interval from first dose date of MMB to death from any cause
Time Frame: Baseline up to the Date of Death or Censoring, up to 3 years
Population: All Enrolled Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5
Number analyzed (Participants) | 7 | 4 | 7 | 3 | 4
Months | 12.4 [3.9 to 22.2] | 5.1 [3.7 to 11.3] | 8.7 [7.3 to 18.3] | 5.6 [4.8 to 18.1] | 7.1 [5.9 to 12.0]

4. Secondary Outcome: Lead-In Phase: Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time interval from the first dose of MMB to the earlier of the first documentation of definitive disease progression or death from any cause. Definitive disease progression is progression based on Response Evaluation Criteria In Solid Tumors (RECIST) criteria v1.1. Data from survival, non-progressing participants will be censored at the earliest of the time of initiation of anti-tumor therapy other than the study treatment or the last time that lack of definitive disease progression was objectively documented while on study.
Time Frame: Baseline up to the Date of Event or Censoring, up to 3 years
Population: All Enrolled Analysis Set
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5
Number analyzed (Participants) | 7 | 4 | 7 | 3 | 4
Months | 5.3 [1.4 to 7.4] | 3.2 [1.9 to 4.8] | 5.5 [5.3 to 7.2] | 5.3 [0.0 to 13.0] | 5.5 [4.5 to 10.1]

5. Secondary Outcome: Lead-In Phase: Overall Response Rate (ORR)
Description: The ORR was defined as the proportion of participants who achieved a best overall response (BOR) during MMB therapy of complete response (CR) or partial response (PR) as assessed by RECIST v1.1.
Time Frame: Baseline up to the Last Tumor Assessment Date, up to 3 years
Population: All Enrolled Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5
Number analyzed (Participants) | 7 | 4 | 7 | 3 | 4
Participants
  Complete Response (CR) | 2 | 1 | 3 | 1 | 0
  Partial Response (PR) | 2 | 2 | 4 | 1 | 4

6. Secondary Outcome: Randomized Treatment Phase: Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time interval from the first dose of MMB to the earlier of the first documentation of definitive disease progression or death from any cause
Time Frame: Baseline up to the Date of Event or Censoring, up to 3 years
Population: The study was discontinued before initiation of the randomized treatment phase.
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Randomized Treatment Phase: Overall Response Rate
Description: The ORR was defined as the proportion of subjects who achieved a best overall response (BOR) during MMB therapy of complete response (CR) or partial response (PR)
Time Frame: Baseline up to the Last Tumor Assessment Date, up to 3 years
Population: The study was discontinued before initiation of the randomized treatment phase.
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (maximum exposure= 63.7 weeks)
Description: Safety Analysis Set: all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | MMB Dose Level 1 | MMB Dose Level 2 | MMB Dose Level 3 | MMB Dose Level 4 | MMB Dose Level 5
All-Cause Mortality (participants affected / at risk) | 4/7 | 3/4 | 6/7 | 0/3 | 3/4
Serious Adverse Events (participants affected / at risk) | 4/7 | 3/7 | 5/7 | 2/3 | 4/4
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4 | 7/7 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMB Dose Level 1 (N=7) | MMB Dose Level 2 (N=7) | MMB Dose Level 3 (N=7) | MMB Dose Level 4 (N=3) | MMB Dose Level 5 (N=4)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MMB Dose Level 1 (N=7) | MMB Dose Level 2 (N=4) | MMB Dose Level 3 (N=7) | MMB Dose Level 4 (N=3) | MMB Dose Level 5 (N=4)
Anaemia (Blood and lymphatic system disorders) | 6 | 2 | 4 | 2 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Intracardiac mass (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 3 | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 3 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3 | 3 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 4 | 4 | 3 | 3
Pancreatic failure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 4 | 0 | 3
Asthenia (General disorders) | 1 | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 2 | 1 | 0
Early satiety (General disorders) | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 3 | 6 | 2 | 4
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1 | 1 | 0
Malaise (General disorders) | 1 | 2 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 4 | 1 | 2 | 2 | 3
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 2 | 3 | 1 | 3
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 3 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 3 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 1 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 1 | 1 | 1
Platelet count decreased (Investigations) | 1 | 0 | 2 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 2 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 2 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 3 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Dizziness exertional (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 0 | 3 | 2 | 2
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 3 | 2 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1 | 2 | 2 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 2 | 1 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Personality change (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 1
Embolism venous (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 2 | 2 | 3
Hypotension (Vascular disorders) | 1 | 0 | 2 | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Sierra Oncology, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Sierra Oncology in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Study Protocol: Original (2014-02-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT02101021/Prot_005.pdf
  • Study Protocol: Amendment 1 (2014-03-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02101021/Prot_006.pdf
  • Study Protocol: Amendment 2 (2014-08-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT02101021/Prot_007.pdf
  • Study Protocol: Amendment 3 (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT02101021/Prot_008.pdf
  • Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT02101021/SAP_009.pdf